CLINICAL TRIAL: NCT02334189
Title: Targeted Letters to Reduce Avoidable Emergency Department Attendances
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Behavioural Insights Team (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2014055
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Avoidable Emergency Department Attendances
MeSH Terms: interventions — College Fraternities and Sororities

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Letter (Experimental): Patients receive a letter containing information on alternative healthcare options for non-emergency health concerns.
  Interventions: Behavioral: Letter
- No letter (No Intervention): Patients receive no letter (this is the usual care).

INTERVENTIONS:
Behavioral: Letter — Patients receive an information letter following an avoidable visit to the Emergency Department.
  Arms: Letter

SUMMARY:
The study aims to test whether it is possible to reduce pressure on Emergency Departments by sending a personal feedback letter to people who have recently attended an Emergency Department and whose health issues could likely have been dealt with elsewhere. These attendances clearly have many causes. However, it is likely that some attendances are due to behavioural factors - in other words, the various ways in which users interact with services. This study focuses on one particular behavioural factor: lack of feedback to users making avoidable visits.

The study will take place in collaboration with an NHS hospital trust. Each week during the trial, the hospital trust will identify those Emergency Department attendances in the last seven days which, according to clinical judgement, could have been dealt with elsewhere. Patients will then be randomly selected to receive a letter containing information on alternative healthcare options for non-emergency health concerns. Patient records will be analysed to determine whether the patients who received the letter are less likely to make an avoidable repeat visit to the Emergency Department in the future, compared with patients who received no letter.

ELIGIBILITY:
Inclusion Criteria:

* Adults who attended a participating Emergency Department during the trial period and whose attendance was codes as 'No Investigation No Significant Treatment'

Exclusion Criteria:

* Children under the age of 18
* All departments and hospitals other than participating Emergency Departments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25000 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Number of avoidable Emergency Department re-attendances (Attendances are classified as avoidable using the 'No Investigation No Significant Treatment' code.) | Measured at 4 months after previous attendance
  Attendances are classified as avoidable using the 'No Investigation No Significant Treatment' code.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Behrendt, MPhil, BA, Principal Investigator — Behavioural Insights Team